CLINICAL TRIAL: NCT07221890
Title: A Trial of Academic Detailing to Promote Prescribing of Biosimilars
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Humana Healthcare Research, Inc. (Unknown)
Responsible Party: Principal Investigator, Benjamin Rome, Assistant Professor of Medicine, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2025P002143
Record Dates: First submitted 2025-10-24; First posted 2025-10-28 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Autoimmune Diseases; Rheumatoid Arthritis (RA); Inflammatory Bowel Disease (IBD); Psoriasis (PsO)
Keywords: biosimilar; biologic; academic detailing; clinician education; prescribing; Medicare Part D
MeSH Terms: conditions — Autoimmune Diseases; Arthritis, Rheumatoid; Inflammatory Bowel Diseases; Psoriasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Offered an academic detailing session either in-person or virtually (depending on assigned geographic region), plus standard-of-care outreach from the insurance plan.
  Interventions: Other: Offered an academic detailing session; Other: Standard-of-care outreach from the insurance plan
- Control (Active Comparator): Not offered an academic detailing session. Standard-of-care outreach from the insurance plan.
  Interventions: Other: Standard-of-care outreach from the insurance plan

INTERVENTIONS:
Other: Offered an academic detailing session — Clinicians will be offered an academic detailing session that will be delivered by a specially trained pharmacist, nurse, or physician (i.e., detailer). These academic detailers will be provided and trained by an independent non-profit organization. After a clinician agrees to participate in an academic detailing session, the detailer will schedule a 1-on-1 meeting lasting 15-20 minutes during which the detailer will provide educational information about biosimilars tailored to their knowledge and attitudes on the topic. During the session, the clinician will be provided printed and/or digital materials, including an educational brochure and patient education materials. Clinicians will also receive access to a summary evidence document containing all of the material with citations. Clinicians will also be offered the opportunity to claim continuing medical education (CME) credits for participating.
  Arms: Intervention
Other: Standard-of-care outreach from the insurance plan — Clinicians will receive formulary information from Humana to provide information about coverage of adalimumab (Humira) and its biosimilars.

SUMMARY:
The goal of this trial is to learn if an interactive evidence-based educational outreach visits to clinicians who prescribe biologics change prescribing of biosimilar medications. The main questions it aims to answer are:

1. Do educational outreach visits lead to a higher number of prescriptions for biosimilar versions of adalimumab?
2. Do in-person or virtual visits work better?

Researchers will compare clinicians offered the educational outreach visit to those who are not offered the visit to see if there is a difference in prescribing of biosimilar versions of adalimumab instead of the original brand-name version.

Participants will be offered the chance to meet with a trained clinician who will provide educational information tailored to their knowledge and attitudes on the topic. They will also be provided an educational brochure and patient educational materials.

DETAILED DESCRIPTION:
This is a parallel, cluster randomized controlled trial in which medical practices with clinicians who prescribed adalimumab (Humira) to patients in a Humana Medicare Prescription Drug Plan (PDP) will be randomized to have eligible clinicians within the practice invited to participate in the educational module about biosimilars (the intervention group). Practices with eligible physicians that are not offered the educational module will serve as the comparison group (the control group). The study will include practices in all 50 US states and Washington, DC, and practices will be stratified into approximately 50 geographic regions. Regions containing about half of the eligible clinicians will have the module offered to the intervention group in-person and the other half of regions will have the module offered virtually. Practices will be randomized 2:1 to be offered detailing (intervention) vs. not be offered detailing (control). Outcomes, including the use and cost of biologics and biosimilars, will be measured from routinely-collected prescribing data using the Humana Research Database.

ELIGIBILITY:
Inclusion Criteria:

* Wrote 7 or more adalimumab prescriptions that were filled by patients enrolled in research-eligible Humana Medicare Part D plans in the calendar year 2025

Exclusion Criteria:

* Retired
* Not able to identify active clinical practice in the US (50 states plus Washington DC)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1325 (Estimated)
Dates: Start 2025-11-06 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Number of biosimilar adalimumab prescriptions per clinician | 12 months
Number of originator adalimumab (Humira) prescriptions per clinician | 12 months
Total spending (payer + patient) on adalimumab | 12 months
Patient out-of-pocket spending on adalimumab | 12 months

SECONDARY OUTCOMES:
Number of participants in the intervention arm who participated in an educational meeting with an academic detailer | 6 months
Number of filled biosimilar prescriptions for other medications with biosimilar versions available, including ustekinumab, tocilizumab, and infliximab | 12 months
Number of filled prescriptions for other brand-name disease-modifying medications that are FDA approved to treat 1 or more of the same indications as adalimumab, such as TNF-alpha inhibitors and interleukin inhibitors | 12 months
Number of patients who fill 1 or more prescriptions for biosimilar adalimumab who subsequently switch back to originator biologic | 12 months

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Humana Healthcare Research, Inc., Louisville, Kentucky
  - Brigham and Women's Hospital, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Undecided
Depends on data use agreement with Humana.